CLINICAL TRIAL: NCT05442320
Title: Influence of Different Toothpaste on Fluoride Concentration in Nails and Dental Fluorosis
Brief Title: Nails and Teeth as Biomarkers of Fluoride Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NAIL1
Record Dates: First submitted 2021-12-03; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2021-12

CONDITIONS: Fluorosis, Dental
Keywords: Dental fluorosis; Fingernails fluoride concentration; Fluoride toothpaste concentration
MeSH Terms: conditions — Fluorosis, Dental

STUDY DESIGN:
Intervention Model Description: Two parallel groups with different toothpaste fluoride concentrations (500 ppm, 1000 ppm)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Same packages of toothpastes with different concentration Key known only to principal investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 500 ppm (Active Comparator): Toothpaste with 500 ppm fluoride (Biodent, Ilirija d.d)
  Interventions: Device: Biodent Toothpaste (Ilirija d.d., Ljubljana, Slovenia)
- 1000 ppm (Experimental): Toothpaste with 1000 ppm fluoride (Biodent, Ilirija d.d)
  Interventions: Device: Biodent Toothpaste (Ilirija d.d., Ljubljana, Slovenia)

INTERVENTIONS:
Device: Biodent Toothpaste (Ilirija d.d., Ljubljana, Slovenia) — Toothpaste with 500 or 1000 ppm of fluoride

SUMMARY:
To determine fluoride concentration in fingernails and estimate if there is a correlation between fluoride concentration in fingernails and fluoride concentration in toothpaste used. In addition, fluorosis of permanent incisors will be evaluated at 13 years of age and correlated with toothpaste fluoride concentration.

DETAILED DESCRIPTION:
Toothpaste with 1000 ppm fluoride and above are more effective in a caries prevention in comparison to toothpastes with lower fluoride concentration or to placebo. Higher fluoride concentrations in toothpastes increase risk for development of tooth fluorosis. Children in first three years of life are most susceptible due to formation of permanent incisors and first molars in this period, beside younger children ingest more toothpaste compared to older children. Fluoride exposure can be measured in nails, where the average plasma fluoride concentration is reflected. The aim of our study was to determine fluoride concentration in fingernails and estimate if there is a correlation between fluoride concentration in fingernails and fluoride concentration in toothpaste used. In our study were included parents and children who had participated in previous studies from parenting class until children's 3 years of age. At that time children were randomly assigned to one of two groups, of which one was being given a toothpaste with 500 ppm fluoride and the other with 1000 ppm fluoride. Children were examined regularly until the age of 3. Children were invited to participate in another clinical examination at 4 years of age. At the time of examination parents were asked to fulfil a questionnaire about oral hygiene habits and a sample of children's fingernails were taken. A questionnaire fulfilled 200 parents, 169 children were examined, finger nail fluoride was analysed by using a gas chromatography method in 161 children. We determined that in 76 % the toothpaste chosen was not appropriate according to EAPD guidelines, 66 % parents was using toothpaste with 500 ppm fluoride for their children. The mean fingernail concentration was 1,43 ng/mg (SD = 0,08). The difference between groups using toothpastes with different fluoride concentrations, and compared with other factors, was not statistically significant. The mean concentration of fluoride in nails of our test group was low compared to reported values in similar studies and there was no significant difference between groups regarding to toothpaste used.

In addition, fluorosis of permanent incisors will be evaluated at 13 years of age and correlated with toothpaste fluoride concentration.

ELIGIBILITY:
Inclusion Criteria:

* participation in parenting class
* normal pregnancy

Exclusion Criteria:

* chronic systemic diseases
* genetic conditions
* complications at delivery

Ages: 0 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 342 (Actual)
Dates: Start 2010-01-03 (Actual); Primary Completion 2014-03-05 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Dental fluorosis | 6 years after permanent incisor eruption
  Dean index

SECONDARY OUTCOMES:
Fingernails fluoride concentration | 4 years of age
  ng/mg

OTHER OUTCOMES:
Caries in primary dentition | 4 years of age
  ICDAS

IPD SHARING:
Plan to Share IPD: Undecided